CLINICAL TRIAL: NCT00500084
Title: An Open-Label Clinical Study Evaluating the Long Term Safety of ALTU-135 in the Treatment of Patients With Exocrine Pancreatic Insufficiency Due to Chronic Pancreatitis or Pancreatectomy
Brief Title: Phase III ALTU-135 CP Safety Trial
Acronym: DIGEST CP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14294; I5L-MC-TCAD (Other: Eli Lilly and Company); 810 (Other: Altus/Alnara)
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Exocrine Pancreatic Insufficiency
Keywords: Chronic Pancreatitis; Pancreatectomy
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis, Chronic | interventions — liprotamase lipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liprotamase (Experimental): Liprotamase is a fixed combination of lipase (32,500 units), protease (25,000 units) and amylase (3,750 units) administered orally with each of three meals and two snacks daily for 12 months
  Interventions: Drug: Liprotamase

INTERVENTIONS:
Drug: Liprotamase — Administered orally
  Other Names: ALTU-135; LY3031642; TheraCLEC - Total

SUMMARY:
This is an open-label, single-arm clinical study investigating the long-term safety of ALTU-135 treatment in Chronic Pancreatitis (CP) patients with exocrine Pancreatic Insufficiency (PI).

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential must be willing to use birth control
* Fecal elastase levels < 100 micrograms per gram (µg/g) stool measured at screening
* Able to perform the testing and procedures required for the study, as judged by the investigator
* Diagnosis of chronic pancreatitis or status post pancreatectomy

Diagnosis of chronic pancreatitis is based upon at least one of the following:

* Endoscopic retrograde pancreatography, magnetic resonance cholangiopancreatography (MRCP) or endoscopic ultrasound demonstrating ductal changes consistent with chronic pancreatitis
* Abnormal Secretin Pancreatic Function test with a peak bicarbonate concentration < 75 milliequivalents per liter (mEq/L)
* Presence of pathognomic pancreatic calcifications
* Pathology proven chronic pancreatitis on surgical specimens

Exclusion Criteria:

* Pregnancy, breastfeeding or of childbearing potential and not willing to use methods of birth control during the study
* History of liver transplant
* Liver transaminases >3x Upper Limit Normal (ULN) or total bilirubin >1.5x ULN at screening or at Baseline (except for patients with Gilbert's Syndrome)
* Participation in an investigational study of a drug, biologic, or device not currently approved for marketing within 30 days prior to screening
* Any condition that the investigator believes would interfere with the intent of this study or would make participation not in the best interest of the patient
* History of pancreatic cancer
* Diagnosis of cystic fibrosis
* Active alcohol or drug abuse
* Presence of any medical condition that is likely to preclude survival for 12 months
* Demonstrated unlikely to comply with protocol requirements or complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with an adverse event | Baseline up to 12 months

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamden, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lebanon, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mineola, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio